CLINICAL TRIAL: NCT05861778
Title: An Open-label, Phase I Study to Evaluate the Safety, Radiation Dosimetry and Pharmacokinetics of 89Zr-TLX250 PET/CT in Patients With Indeterminate Renal Masses or Suspected Recurrent Renal Clear Cell Carcinoma
Brief Title: Evaluation of 89Zr-TLX250 PET/CT in Chinese Patients With Indeterminate Renal Masses or Suspected Recurrent Renal Clear Cell Carcinoma
Acronym: ZIRDOSE-CP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Collaborators: Grand Pharmaceutical (China) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TLX250CDx-CP-001
Record Dates: First submitted 2023-04-05; First posted 2023-05-17 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Clear Cell Renal Cell Carcinoma; Suspected Recurrent Renal Clear Cell Carcinoma; Recurrent Renal Cell Cancer
Keywords: indeterminate renal masses; Suspected Recurrent Renal Clear Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-girentuximab (Experimental): A single administration of 37 MBq (+/-10%) 89Zr-girentuximab, containing a mass dose of 10 mg of girentuximab
  Interventions: Drug: 89Zr-Girentuximab

INTERVENTIONS:
Drug: 89Zr-Girentuximab — A single administration of 37 MBq (±10%) 89Zr-TLX250, containing a mass dose of 10 mg of girentuximab, followed by whole body PET/CT scans were performed at 0.5h, 4h, 24h, 72 hours and 7±1 days post administration.
  Other Names: 89Zr-DFO-girentuximab; 89Zr-TLX250; TLX250CDx

SUMMARY:
The study is designed to evaluate the safety, tolerability, radiation dosimetry and pharmacokinetics 89Zr-TLX250 (also known as 89Zr-DFO-girentuximab) Positron Emission Tomography/Computed Tomography (PET/CT) in adult Chinese patients with indeterminate renal masses or Suspected Recurrent Renal Clear Cell Carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed written informed consent
2. Chinese male or female≥18 years old.
3. Have an indeterminate renal mass, suspected renal cell carcinoma, or previously diagnosed ccRCC, suspected recurrence on the pre-screening imaging from Day -90 to Day -1
4. Negative serum pregnancy test for female subjects of childbearing potential at screening. Confirmed negative urine pregnancy test within 24 hours prior to administration of investigational product.
5. Expected survival ≥ 6 months.
6. Agree to follow appropriate and highly effective contraception method for at least 35 days after the administration of 89Zr-TLX250.

Exclusion Criteria:

1. Renal mass is known to be a metastasis of another primary tumor.
2. Have other malignancies that require treatment.
3. Planned antineoplastic therapies (for the period between IV administration of 89Zr-TLX250 and imaging).
4. Have received chemotherapy, radiotherapy, or immunotherapy within 4 weeks prior to the planned administration of 89Zr-TLX250 or such therapy resulted in a persistent adverse event (> Grade 1) (per National Cancer Institute-Common Toxicity Criteria version 5.0 [NCICTCAE v5.0]).
5. Exposure to murine or chimeric antibodies within the last 5 years.
6. Prior use of radionuclides with an interval of less than 10 halflives.
7. Exposure to any investigational diagnostic or therapeutic agent within the first 4 weeks or 5 half-lives (whichever is longer) of the planned administration of 89Zr-TLX250.
8. Renal insufficiency with glomerular filtration rate (GFR) ≤ 60 mL/min/1.73 m².
9. Uncontrolled psychiatric disorders.
10. Women who are pregnant or breastfeeding.
11. Known hypersensitivity to girentuximab or DFO (deferoxamine).
12. Have a serious non-malignant disease (e.g., infectious disease, autoimmune disease, or metabolic disease) that, in the opinion of the investigator, may interfere with the purpose of the study or subject safety or compliance.
13. Vulnerable population (e.g., being in detention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Safety parameter Physical Examination | 9 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding the physical examination.
Safety parameter Vital Signs | 9 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding the Vital signs
Safety parameter Laboratory examinations | 9 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding Laboratory examinations.
Safety parameter concomitant medications | 9 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding concomitant medications.
Safety parameter ECG | 9 days
  Frequency of occurrence and severity of abnormal findings in the 12-lead ECG (ECG QT Interval)

SECONDARY OUTCOMES:
Whole blood radioactivity PK parameters | 6 days
  This outcome will be measured by analysing the radioactivity present in the blood at baseline (pre-dose), 0.5h, 1h, 2h, 4h, 24h, 72h and Day 5+/-1 day. Assessments include: Cmax (maximum concentration)
Radiation dosimetry | 8 days
  whole body PET/CT scans will be acquired in supine position at 0.5, 4, 24, 72 and 168±24 h (Day 7±1) post injection, using low dose CT without contrast agent. Normalized Absorbed Dose = Absorbed Dose/ Administered Dose
Tumour dosimetry | Whole body PET/CT scans will be acquired in supine position at 0.5, 4, 24, 72 and 168±24 h (Day 7±1) post injection
  Normalised whole body effective radiation dose (mSv/MBq)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Yang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: No